CLINICAL TRIAL: NCT05160974
Title: QTERN (SAXAGLIPTIN/DAPAGLIFLOZIN FDC) Regulatory Post-Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1683R00008
Record Dates: First submitted 2021-11-04; First posted 2021-12-16 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This is a local, prospective, non-interventional, regulatory post-marketing surveillance study. Adult patients with type 2 diabetes mellitus who are initiating Qtern as indicated by the MFDS will be included. 600 patients are followed up 12 weeks and at least 60 patients of the 600 patients are followed up 24 weeks. Patients will be treated as part of routine practice at Korean healthcare centers by accredited physicians. In this study, patients will receive Qtern as indicated in the locally approved prescribing information.

DETAILED DESCRIPTION:
As part of a post approval commitment, the MFDS has requested a post-marketing surveillance program to characterize safety in patients who are treated with Qtern for T2DM by physicians in the normal clinical practice setting. This study is designed to confirm assess the known safety profile or identify previously unsuspected adverse reactions and to evaluate the effectiveness of Qtern under conditions of routine daily medical practice in Korea.

The primary objective of this study is :

Descriptive analysis of the proportion of adverse events (AEs) and serious adverse events (SAEs) in patients who are treated with Qtern for type 2 diabetes mellitus by physicians in the normal clinical practice setting over a period of 12 and 24 weeks.

The secondary objectives of this study are:

To follow the changes of the hemoglobin A1c (HbA1c), fasting plasma glucose (FPG), 2-hr post-prandial glucose (PPG-2hr), blood pressure, abdominal circumference and body weight and self-reported data in this cohort of patients from baseline to completion of the study.

To evaluate the safety and tolerability of Qtern in patients with type 2 diabetes mellitus based on conducted laboratory test. (Laboratory tests are not mandatory because of the non-interventional nature of this study)

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years and older
2. Patients with T2DM eligible for treatment with Qtern as indicated in the locally approved prescribing information
3. Patients with evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Patients treated with Qtern outside of the locally approved Prescription Information in Korea
2. Patients with contraindications for the use of Qtern (as described in the Korean Prescription Information)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are diagnosed with T2DM eligible for the treatment with Qtern (5 mg saxagliptin/10 mg dapagliflozin) according to prescription information approved by MFDS and as decided by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
• Incidence (%) of AEs in patients who are treated with Qtern | 12 or 24 weeks
• Nature of AE in patients who are treated with Qtern | 12 or 24 weeks
• Nature of unexpected adverse drug reactions in patients who are treated with Qtern | 12 or 24 weeks
• Severity of AE in patients who are treated with Qtern | 12 or 24 weeks
• Incidence of unexpected adverse drug reactions in patients who are treated with Qtern | 12 or 24 weeks
• Severity of unexpected adverse drug reactions in patients who are treated with Qtern | 12 or 24 weeks
• Incidence (%) of SAEs in patients who are treated with Qtern | 12 or 24 weeks

SECONDARY OUTCOMES:
• Change in HbA1c during the observation period | 12 or 24 weeks
• Change in FPG during the observation period | 12 or 24 weeks
• Change of PPG-2hr during the observation period | 12 or 24 weeks
• Change in blood pressure during the observation period | 12 or 24 weeks
• Change in abdominal circumference during the observation period | 12 or 24 weeks
• Change in body weight during the observation period | 12 or 24 weeks
• Overall assessment on the outcome of the treatment by investigators | 12 or 24 weeks
  The overall investigator's assessment on the outcome will be based on the investigator's clinical judgment and classified as below criteria issued by the Korean Ministry of Food and Drug Safety (MFDS):
  * Improved: Signs and symptoms are significantly improved or maintenance effect
  * Unchanged: Improvement in signs and symptoms is not significant or there is no change in signs and symptoms
  * Worsened: Signs and symptoms are worsened
  * Assessment impossible: Assessment is impossible because the surveillance drug was discontinued before 12 weeks
• Clinically significant results from blood chemistry test | 12 or 24 weeks
  Clinically significance will be determined as per the investigators clinical judgement based on routine clinical practice.
• Clinically significant results from complete blood count test | 12 or 24 weeks
  Clinically significance will be determined as per the investigators clinical judgement based on routine clinical practice.
• Clinically significant results from urinalysis | 12 or 24 weeks
  Clinically significance will be determined as per the investigators clinical judgement based on routine clinical practice.

CONTACTS AND LOCATIONS:
Locations (23):
- South Korea (23):
  - Research Site, Changwon-si, South Korea
  - Research Site, Gimcheon, South Korea
  - Research Site, Jeju-do, South Korea
  - Research Site, Jeonju, South Korea
  - Research Site, Pyeongtaek-si, South Korea
  - Research Site, Seosan City, South Korea
  - Research Site, Yeongcheon-si, South Korea
  - Research Site, Busan
  - Research Site, Changwon
  - Research Site, Cheongju-si
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Gwangju
  - Research Site, Gwangmyeong
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Jeonju
  - Research Site, Jinju
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan
  - Research Site, Yongin-si

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D168300008_Study Report Synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1683R00008&attachmentIdentifier=7010e16d-d7bf-4220-9583-8c6a8e5b68b2&fileName=D168300008_Study_Report_Synopsis_2.0_redacted.pdf&versionIdentifier=